CLINICAL TRIAL: NCT01080313
Title: Prospective, Longitudinal, Multi-Center, Descriptive Registry of Patients Receiving Therapy Other Than Surgical Resection Alone for Newly Diagnosed Head and Neck Cancer
Brief Title: Head and Neck Cancer Registry (LORHAN)
Acronym: LORHAN
Status: Completed | Type: Observational
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 13440; I4E-US-S003 (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-03-02; First posted 2010-03-04 (Estimated); Last update posted 2012-02-13 (Estimated); Status verified 2012-02

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Therapeutics

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with head and neck cancer
  Interventions: Other: Therapy for head and neck cancer

INTERVENTIONS:
Other: Therapy for head and neck cancer — radiotherapy and/or drug therapy including chemotherapy, biologic therapy and targeted therapy

SUMMARY:
The primary objective of this study is to describe, in detail, patterns of care for head and neck carcinoma patient

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) confirmed new diagnosis of carcinoma involving the oral cavity, oropharynx, nasopharynx, hypopharynx, larynx, or neck node metastasis from unknown origin
* Scheduled to receive radiotherapy and/or drug therapy including chemotherapy, biologic therapy and targeted therapy
* Written informed consent

Exclusion Criteria:

* Registry participation does not exclude participation in clinical trials.
* Patients scheduled to receive or who have received surgery are eligible for Registry participation as long as they are also scheduled to receive medical therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 26000 (Estimated)
Dates: Start 2005-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Patterns of care for head and neck cancer | up to 10 years

SECONDARY OUTCOMES:
Overall survival by treatment regimen | study entry to death from any cause or to end of study
Determine the incidence and severity of major dose-limiting and other important treatment toxicities | up to 10 years
Identify supportive care received for managing nutrition, pain, nausea and other complications | up to 10 years
tumor control by treatment regimen | study entry to progressive disease

CONTACTS AND LOCATIONS:
Overall Officials: Mednet Solutions, Study Director — MedNet Solutions
Locations (1):
- Mednet Solutions, Minnetonka, Minnesota, United States